CLINICAL TRIAL: NCT00226811
Title: An Open Label International Multi-Center Phase 2 Activity And Safety Study Of SU011248 In Patients With Advanced / Metastatic Gastric Cancer Progressing Or Recurring After One Prior Chemotherapy
Brief Title: An International Phase 2 Study Of SU011248 In Patients With Advanced / Metastatic Gastric Cancer Failing Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181054
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Results first posted 2009-11-26 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): 50mg daily, taken by mouth for 28 days followed by 2 weeks of drug free period was one cycle. Cycles were repeated until progression of disease or unacceptable toxicity was observed
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — 50mg daily, taken by mouth for 28 days followed by 2 weeks of drug free period was one cycle. Cycles were repeated until progression of disease or unacceptable toxicity was observed

SUMMARY:
The study consisted of two parts. In Part 1 the study enrolled 38 patients (Step 1 Simon 2 step design) after which Step 2 was opened and the total enrollment target for the study (n=63) was exceeded due to a rapid enrollment (78 patients were entered). Part 2 of the study did not open due to the final overall insufficiency of efficacy observed in 78 patients. Sunitinib (SU011248) was administered orally daily for 4 weeks followed by a 2-week rest at a starting dose of 50 mg with provision for dose reduction based on tolerability. All patients received repeated cycles of sunitinib until disease progression, occurrence of unacceptable toxicity, or other withdrawal criteria were met. After discontinuation of treatment, patients were followed up in order to collect information on further antineoplastic therapy and survival.

ELIGIBILITY:
Inclusion Criteria:

* Gastric or gastroesophageal junction adenocarcinoma cyto/histologically documented
* Disease progression/ recurrence after treatment with one prior single agent or combination chemotherapy regimen for advanced / metastatic disease (last dose at least 4 wks before study entry). Patients may have also received prior adjuvant therapy if recurrence occurred > 6 months after adjuvant therapy completion
* Evidence of measurable disease by radiographic technique
* Adequate organ function.

Exclusion Criteria:

* Clinically relevant ascites (i.e. requiring paracentesis)
* Severe weight loss
* NCI CTCAE Grade 3 hemorrhage <4 weeks of starting study treatment
* Diagnosis of second malignancy within last 3 years
* History of or known brain metastases, spinal cord compression, or carcinomatous meningitis
* Known HIV
* Serious acute or chronic illness
* Current treatment on another clinical trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- China (3):
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Guangzhou
- Hong Kong (2):
  - Pfizer Investigational Site, Hong Kong
  - Pfizer Investigational Site, Shatin
- Italy (2):
  - Pfizer Investigational Site, Ancona
  - Pfizer Investigational Site, Genova
- Japan (3):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Suntougun, Shizuoka
  - Pfizer Investigational Site, Chuo-ku, Tokyo
- Pfizer Investigational Site, Porto, Portugal
- Pfizer Investigational Site, Seoul, South Korea
- Taiwan (2):
  - Pfizer Investigational Site, Kwei-Shan, Taoyuan
  - Pfizer Investigational Site, Taipei

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181054&StudyName=An%20International%20Phase%202%20Study%20Of%20SU011248%20In%20Patients%20With%20Advanced%20/%20Metastatic%20Gastric%20Cancer%20Failing%20Chemotherapy

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study used a Simon 2-stage design with objective response rate (ORR) as the primary efficacy endpoint. Enrollment was halted after Part 1 Stage 2 because the minimum number of responding subjects required to proceed to Part 2 was not reached. Further subject enrollment therefore ended after 78 subjects had been enrolled and treated on Part 1.
Groups:
- 50 mg Sunitinib: Sunitinib was administered orally daily for 4 weeks followed by a 2-week off-treatment period (Schedule 4 weeks on drug / 2 weeks off) in each cycle. The starting dose was 50 mg daily with provision for dose interruption and/or reduction based on tolerability. All subjects received repeated cycles of sunitinib until disease progression, occurrence of unacceptable toxicity, withdrawal of subject consent, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | 50 mg Sunitinib
Started | 78
Completed | 2
Not Completed | 76
Not completed — Death | 8
Not completed — Adverse Event | 11
Not completed — Lack of Efficacy | 55
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 56

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Number of patients with best overall response = complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses were those that persisted on repeat imaging study ≥4 weeks after initial documentation of response. CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From start of study treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: Intent-to-treat (ITT) population includes all patients enrolled in the study that received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 25
  Progressive Disease | 42
  Not Evaluable | 5
  Missing | 4

2. Secondary Outcome: Clinical Benefit Response (CBR)-Complete Response (CR), Partial Response (PR) or Stable Disease (SD) With Duration ≥ 24 Weeks
Description: Number of patients with Clinical Benefit Response: confirmed CR, confirmed PR or stable disease (SD) for at least 24 weeks on study according to the Response Evaluation Criteria in Solid Tumors (RECIST). CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions. SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progessive disease (PD) taking as a reference the smallest sum of the longest dimensions since the treatment started.
Time Frame: From start of study treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or clinical benefit response for at least 24 weeks on study
Population: ITT population
Measure: Number; unit: participants
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
participants | 6
Statistical Analysis 1: Comparison: 50 mg Sunitinib; Test type: Superiority or Other; CBR rate (percentage) = 7.7, 95% CI [2.9 to 16.0] — Clinical benefit response rate: percent of patients with confirmed complete response, confirmed partial response or stable disease for at least 24 wks according to Response Evaluation Criteria in Solid Tumors, relative to total treated patients

3. Secondary Outcome: Duration of Response (CR or PR)
Description: Time from the first documentation of confirmed objective response (CR or PR) to the first documentation of disease progression or to death due to any cause. CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Day 28 of Cycle 1 and Day 28 of Cycles thereafter or death due to cancer
Population: ITT population
Measure: Mean (Full Range); unit: weeks
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 2
weeks | 16 [6 to 26]

4. Secondary Outcome: Progression-Free Survival
Description: Time from start of study treatment to first documentation of objective tumor progression, or to death due to any cause. PFS was calculated as (first event date minus the date of first dose plus 1) divided by 7.
Time Frame: From start of study treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter or death
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
weeks | 10.0 [6.9 to 11.1]

5. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Time from the start of study treatment to the first documentation of objective tumor progression. TTP was calculated as (first event date minus the date of first dose plus 1) divided by 7.
Time Frame: From start of study treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
weeks | 10.1 [7.29 to 11.29]

6. Secondary Outcome: Overall Survival
Description: Time from the date of first dose of study medication to the date of death due to any cause. OS was calculated as (date of death minus the date of first dose date plus 1) divided by 7.
Time Frame: From start of study treatment until death
Population: ITT population
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
weeks | 29.6 [19.1 to 42.0]

7. Primary Outcome: Objective Response (Complete Response (CR) or Partial Response (PR))
Description: Number of patients with Objective Response (OR): confirmed CR or confirmed PR according to the Response Evaluation Criteria in Solid Tumors (RECIST). CR = the disappearance of all target lesions. PR = a ≥30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: From start of study treatment until Day 28 of Cycle 1, Day 28 of Cycles thereafter
Population: ITT population
Measure: Number; unit: participants
Arm/Group | 50 mg Sunitinib
Number analyzed (Participants) | 78
participants | 2
Statistical Analysis 1: Comparison: 50 mg Sunitinib; Test type: Superiority or Other; OR rate (percentage) = 2.6, 95% CI [0.3 to 9.0] — Percentage of patients with confirmed complete response or confirmed partial response according to the Response Evaluation Criteria in Solid Tumors (RECIST), relative to the total number of treated patients

ADVERSE EVENTS:
Arm/Group | 50 mg Sunitinib
Serious Adverse Events (participants affected / at risk) | 30/78
Other Adverse Events (participants affected / at risk) | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Sunitinib (N=78)
Anaemia (Blood and lymphatic system disorders) | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Cardiac arrest (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Heterophoria (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 2
Salivary gland pain (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Disease progression (General disorders) | 6
Fatigue (General disorders) | 2
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Performance status decreased (General disorders) | 1
Pyrexia (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Brain herniation (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Stent occlusion (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Brain stem haemorrhage (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Hypopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg Sunitinib (N=78)
Anaemia (Blood and lymphatic system disorders) | 30
Leukopenia (Blood and lymphatic system disorders) | 30
Lymphopenia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 45
Abdominal distension (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 20
Abdominal pain upper (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 29
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 11
Gingivitis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 31
Stomatitis (Gastrointestinal disorders) | 28
Vomiting (Gastrointestinal disorders) | 22
Asthenia (General disorders) | 7
Face oedema (General disorders) | 4
Fatigue (General disorders) | 35
Malaise (General disorders) | 4
Mucosal inflammation (General disorders) | 11
Oedema (General disorders) | 7
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 20
Hyperbilirubinaemia (Hepatobiliary disorders) | 13
Nasopharyngitis (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 12
Blood alkaline phosphatase increased (Investigations) | 11
C-reactive protein increased (Investigations) | 5
Red blood cell count decreased (Investigations) | 5
Weight decreased (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 36
Hypoalbuminaemia (Metabolism and nutrition disorders) | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyponatraemia (Metabolism and nutrition disorders) | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 9
Dizziness (Nervous system disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 6
Peripheral sensory neuropathy (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 22
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 14
Skin discolouration (Skin and subcutaneous tissue disorders) | 19
Skin exfoliation (Skin and subcutaneous tissue disorders) | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Yellow skin (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 11
Ascites (Gastrointestinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.